CLINICAL TRIAL: NCT06739980
Title: The ENABLE Study: An Open-Label, Long-Term Safety and Efficacy Study of INZ-701 in Patients With Ectonucleotide Pyrophosphatase/ Phosphodiesterase 1 (ENPP1) Deficiency
Brief Title: The ENABLE Study: Safety and Efficacy Study of INZ-701 in Patients With ENPP1 Deficiency
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not initiated as it is no longer consistent with the Sponsor's development plans.
Sponsor: Inozyme Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INZ701-108
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Ectonucleotide Pyrophosphatase/phosphodiesterase1 Deficiency; Autosomal Recessive Hypophosphatemic Rickets; Generalized Arterial Calcification of Infancy 1
Keywords: Ectonucleotide Pyrophosphatase/Phosphodiesterase1 Deficiency; Hypopyrophosphatemia; ENPP1; Autosomal Recessive Hypophosphatemic Rickets Type 2; ARHR2; Generalized Arterial Calcification of Infancy; GACI
MeSH Terms: conditions — Hypophosphatemic Rickets, Autosomal Recessive, 1; Arterial calcification of infancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- INZ-701 (Experimental): INZ-701 will be administered by SC injection on a once-weekly basis as follows:
  * Study participants from 1 year to <18 years of age will receive a dose of 2.4 mg/kg
  * Study participants ≥18 years and:
  weighing <50 kg or >100 kg will receive a 1.8 mg/kg dose,
  OR
  weighing ≥50 and ≤100 kg will receive a 150 mg dose of INZ-701
  Interventions: Drug: INZ-701

INTERVENTIONS:
Drug: INZ-701 — Recombinant fusion protein that contains the extracellular domains of human ENPP1 coupled with an Fc fragment from an immunoglobulin gamma-1 (IgG1) antibody.
  Other Names: (rhENPP1-Fc).

SUMMARY:
The purpose of Study INZ701-108 (ENABLE) is to assess the safety and efficacy of INZ-701 in patients 1 year of age and older with ENPP1 Deficiency who have not previously received INZ-701 and are not eligible for existing Inozyme-sponsored clinical studies that are still open to enrollment.

DETAILED DESCRIPTION:
INZ-701 is an ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) enzyme replacement therapy in development for the treatment of the ultra-rare genetic disorder, ENPP1 Deficiency.

Study INZ701-108 (ENABLE) is an open-label study to assess the long-term safety and efficacy of INZ-701 in patients 1 year of age and older with ENPP1 Deficiency who have not previously received INZ-701 and are not eligible for an Inozyme-sponsored clinical study that is open to recruitment.

The study will consist of a 30-day Screening Period, followed by an open-label Treatment Period during which all participants will receive once-weekly subcutaneous (SC) doses of INZ-701 and continue treatment through 104 weeks. The dose will be determined by the participant's age and weight.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate must meet all of the following inclusion criteria:

1. Provide written or electronic informed consent after the nature of the study has been explained, and prior to any research-related procedures, per International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP)
2. Provide assent in accordance with local regulations, if <18 years of age
3. Male or female, ≥1 year of age
4. A confirmed postnatal molecular genetic diagnosis of ENPP1 Deficiency with biallelic variants (ie, homozygous or compound heterozygous) performed using assays that meet CE-marked requirements, or from a College of American Pathologists/Clinical Laboratory Improvement Amendments (CAP/CLIA) certified laboratory, or regional equivalent
5. Must have at least one of the following clinical signs and/or symptoms consistent with ENPP1 Deficiency:

   1. ≥1 atraumatic vertebral fracture
   2. ≥2 fractures as an adult (eg, long bones, digits, vertebrae)
   3. For participants <55 years of age, low bone mineral density measured at any of the following sites: lumbar spine, radius, and hip (DXA Z-score less than -1.5)
   4. History of myocardial infarction, unstable angina, transient ischemic attack, or low cardiac output before the age of 40 years
   5. Renal vascular hypertension or other evidence for vascular insufficiency/stenosis
   6. History of rickets or bone deformity
   7. Diagnosis of ossification of the posterior longitudinal ligament
   8. Other clinical signs/symptoms, with approval by Inozyme
6. Fasting plasma PPi concentration of <1400 nM at Screening
7. Serum level of 25-hydroxyvitamin D (25[OH]D) ≥12 ng/mL at Screening (Participants may be rescreened after receiving cholecalciferol treatment.)
8. Women of childbearing potential (WOCBP, as defined in Clinical Trials Coordination Group [CTCG 2024]) must have a negative serum pregnancy test at Screening and must not be breastfeeding
9. Males who are sexually active must agree to use condoms from the period following first dose of INZ-701 through 30 days after the last dose of INZ-701
10. WOCBP and partners of fertile males who are WOCBP must be using or agree to use a highly effective form of contraception (as per CTCG 2024) from at least 1 month before the first dose of INZ-701 through 30 days after the last dose of INZ701 (greater than 5 half-lives of INZ-701)
11. In the opinion of the Investigator, able to complete all aspects of the study

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria will not be eligible to participate:

1. In the opinion of the Investigator, presence of any clinically significant disease or laboratory abnormality not due to ENPP1 Deficiency that may confound interpretation of study results
2. Eligible for another Inozyme sponsored study of INZ-701 treatment that is open for enrollment
3. Receiving prohibited medications
4. Unable or unwilling to discontinue calcitriol or other active forms of vitamin D3 (or analogs) within 7 days prior to Day 1 and/or oral phosphate supplements within 36 hours prior to Day 1
5. Received previous treatment with INZ-701
6. Concurrent participation in another interventional clinical study and/or has received an investigational drug within 5 half-lives or within 4 weeks prior to the first dose of INZ-701, whichever is longer
7. Pregnant, trying to become pregnant, or breastfeeding
8. Male participants trying to father a child

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Plasma Inorganic Pyrophosphate (PPi) concentration through Week 52 | 52 weeks (Baseline through Week 52)
  For each subject, plasma PPi will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.

SECONDARY OUTCOMES:
Change from Baseline in skeletal abnormalities as measured by the Radiographic Global Impression of Change (RGI-C) global score through Week 104 for patients 1 to <13 years | 52 weeks (Baseline through Week 52)
  For each subject, skeletal abnormalities will be measured via RGI-C global scores obtained throughout the study, comparing the subject's baseline value over time.
Change from Baseline in Rickets Severity Score (RSS) total score through Week 104 (measured on all long bones with open growth plates in the knee or wrist) for patients 1 to <13 years | 104 weeks (Baseline through Week 104)
  For each subject, rickets severity score will be measured on all long bones with open growth plates in knees or wrist obtained throughout the study, comparing the subject's baseline value over time.
Change from Baseline in arterial calcification score based on low dose computed tomography (CT) through Week 104 for patients 1 to <18 years | 104 weeks (Baseline through Week 104)
  For each subject, arterial calcification will be measured via low dose computed tomography obtained throughout the study, comparing the subject's baseline value over time.
Change over time in serum biomarkers: Fibroblast growth factor 23 for patients >1 year | 104 weeks (Baseline through Week 104)
  For each subject, various serum biomarkers will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change over time in serum biomarkers: Procollagen type 1 N-terminal propeptide for patients >1 year | 104 weeks (Baseline through Week 104)
  For each subject, various serum biomarkers will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change over time in serum biomarkers: Bone-specific alkaline phosphatase for patients >1 year | 104 weeks (Baseline through Week 104)
  For each subject, various serum biomarkers will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change over time in serum biomarkers: Carboxy terminal cross-linked telopeptide of type I collagen for patients >1 year | 104 weeks (Baseline through Week 104)
  For each subject, various serum biomarkers will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time
Change from Baseline in growth parameters (body weight expressed as Z-score) through Week 104 for patients 1 to <13 years | 104 weeks (Baseline through Week 104)
  For each subject, growth parameters will be measured throughout the study, comparing the subject's baseline value over time.
Change over time in serum biomarkers: Serum phosphate for patients >1 year | 104 weeks (Baseline through Week 104)
  For each subject, various serum biomarkers will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change from Baseline in growth parameters (height/length expressed as Z-score) through Week 104 for patients 1 to <13 years | 104 weeks (Baseline through Week 104)
  For each subject, growth parameters will be measured throughout the study, comparing the subject's baseline value over time.
Change from Baseline over time in growth velocity as measured by height over time through Week 104 for patients 1 to <13 years | 104 weeks (Baseline through Week 104)
  For each subject, growth velocity will be measured via height throughout the study, comparing the subject's baseline value over time.
Change from Baseline in lower extremity angle measurements from radiographic x-rays through Week 104 for patients 1 to <13 years | 104 weeks (Baseline through Week 104)
  For each subject, lower extremity angle will be measured via radiograph x-rays throughout the study, comparing the subject's baseline value over time.
Change from Baseline in audiometric outcomes as measured by hearing tests through Week 104 for patients 1 to <18 years | 104 weeks (Baseline through Week 104)
  For each subject, audiometric outcomes will be measured via hearing tests throughout the study, comparing the subject's baseline value over time.
Change from Baseline in 6 Minute Walk Test (6MWT) for patients >5 years | 104 weeks (Baseline through Week 104)
  For each subject, 6-minute walk test will be measured and assessed throughout the study, comparing the subject's baseline value over time.
Change in Baseline in bone mineral content and bone mineral density Z-score via dual X-ray absorptiometry (DXA) scan through Week 104 for patients ≥13 years | 104 weeks (Baseline through Week 104)
  For each subject, bone mineral content and density will be measured via dual x-ray absorptiometry (DXA) throughout the study, comparing the subject's baseline value over time.
Change from Baseline in age-appropriate motor performance-mobility assessments through Week 104 (Peabody Developmental Motor Scale - third edition [PDMS] for patients 1 to < 5 years | 104 weeks (Baseline through Week 104)
  For each subject, motor performance-mobility assessments will be measured via the Developmental Motor Scale throughout the study, comparing the subject's baseline value over time.
Patient Reported Outcomes (PROs) through Week 104 assessed via Patient-Reported Outcome Measurement Information System (PROMIS) Pediatric - Cognitive Function, Fatigue, Pain Intensity, Pain Interference, Mobility) for patients 1 to <18 years | 104 weeks (Baseline through Week 104)
  For each subject, quality of life PROs will be assessed throughout the study, comparing the subject's baseline value over time.
PROs through Week 104 (Patient-Reported Outcome Measurement Information System [PROMIS] Pediatric - Cognitive Function, Fatigue, Pain Intensity, Pain Interference, Physical Function) for patients >17 years | 104 weeks (Baseline through Week 104)
  For each subject, quality of life PROs will be assessed throughout the study, comparing the subject's baseline value over time.
PROs through Week 104 (Clinical-, Caregiver-, and Patient-reported Global Impression of Change [CGI-C, CaGI-C, and PGI-C for patients >17 years | 104 weeks (Baseline through Week 104)
  For each subject, PROs will be assessed throughout the study, comparing the subject's baseline value over time.
Change from Baseline in bone histomorphometry as measured by bone biopsy through Week 104 for patients >17 years | 104 weeks (Baseline through Week 104)
  For each subject, bone histomorphometry will be measured via bone biopsy throughout the study, comparing the subject's baseline value over time.
Change from Baseline in pain visual analog VAS) score through Week 104 for patients >17 years | 104 weeks (Baseline through Week 104)
  For each subject, pain will be measured via pain visual analog scale throughout the study, comparing the subject's baseline value over time.

OTHER OUTCOMES:
Number of Treatment Adverse Events (TEAEs) through Week 104 | 104 weeks (Baseline through Week 104)
  Treatment-emergent AEs are defined as any AE occurring from the first dose of INZ-701 through 30 days after the last dose of INZ-701.
Incidence of Anti-Drug Antibodies (ADA) through Week 104 | 104 weeks (Baseline through Week 104)
  For each subject, the presence of ADAs will be assessed and, if present, further evaluation will determine specificity and subtypes.

CONTACTS AND LOCATIONS:
Overall Officials: Inozyme Pharma, Inc., Study Director — Inozyme Pharma, Inc.

IPD SHARING:
Plan to Share IPD: No